CLINICAL TRIAL: NCT04151758
Title: Effect of Docosahexaenoic Acid Supplementation on Microbiome in Obese ChiLdrEn. The DAMOCLE Study
Brief Title: Effect of Docosahexaenoic Acid Supplementation on Microbiome in Obese ChiLdrEn.
Acronym: DAMOCLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Elvira Verduci, PhD, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/ST/135-1
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Gut microbiota; Nutrition; PUFA supplementation
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docosahexaenoic Acid Supplementation, lifestyle intervention (Experimental): Docosahexaenoic Acid (DHA) will be given at the dose of 500 mg/day. Physical activity and healthy eating habits will be encouraged.
  Interventions: Drug: Docosahexaenoic Acid Supplementation; Other: Promotion of physical activity; Other: Promotion of healthy food habits

INTERVENTIONS:
Drug: Docosahexaenoic Acid Supplementation — Docosahexaenoic Acid (DHA) will be given at the dose of 500 mg/day (2 ml per day DHA RICH OIL 25% aroma mandorla FoodAR Limbiate, Italy;50% DHA oil obtained from Schyzochitrium sp ; Martek Biosciences Corporation, Columbia, Maryland, USA) to all participants of the study. DHA 2 ml will provide about 16 kcal of energy.
  Other Names: Lifestyle intervention; Diet intervention
Other: Promotion of physical activity — All participants will underwent a visit at t0, t1 and t2 in which physical activity will be promoted according to Italian dietary guidelines for childhood obesity.
Other: Promotion of healthy food habits — All participants will underwent a visit at t0, t1 and t2 in which healthy food habits will be promoted according to Italian dietary guidelines for childhood obesity.

SUMMARY:
Evaluation of the possible effect of DHA supplementation, combined with interventions aimed at improving diet and lifestyle, on gut microbiota composition and metabolite production.

DETAILED DESCRIPTION:
Differences in gut microbiota composition and function will be evaluated in obese children before starting the DHA supplementation and dietary-lifestyle intervention, at the end of DHA supplementation (4 months) e after 4 months of dietary dietary-lifestyle intervention without DHA supplementation. The investigators will identify the role of DHA on the intestinal microbiota and indicative species related to insulin resistance (IR). The investigators will determine whether DHA supplementation, combined with interventions to improve diet and lifestyle, reduces adverse metabolic consequences together with their co-morbidities.

The following tasks will be also performed at t0, t1 and t2:

Clinical examination including: physical examination, Tanner score evaluation; Bristol Stool Chart Blood pressure will be checked in all children by using oscillometric devices validated in the pediatric age group.

Anthropometry including body circumferences and skinfolds, calculation of BMI z scores and body composition. Body composition will be assessed using an air displacement plethysmography system (BOD POD COSMED-USA).

Dietary assessment:

* Food intakes will be recorded by prospective 3-d weighed food records obtained with food scales. Parents will be advised on how to record all food and beverages consumed during 2 weekdays and 1 weekend day. Quantification and analysis of the energy intake and nutrient composition will be performed with an ad hoc PC software (MètaDieta®, Me.Te.Da S.r.l., San Benedetto del Tronto, Italy).
* Mediterranean Diet Quality Index (KIDMED) questionnaire for Mediterranean Diet assessment. The KIDMED index ranges from 0 to 12, and is based on a 16-question test that can be self-administered. The sums of the values from the administered test will be classified into three levels:

  8 or more: optimal Mediterranean diet; 4-7: improvement needed to adjust intake to Mediterranean patterns. 3 or less: very low diet quality.

Hematological and biochemical status including:

Complete cell blood count;

Metabolic and nutritional parameters according to local routines for childhood obesity (fasting glucose, fasting insulin, LDL, HDL, total cholesterol, triglycerides, Apolipoprotein A and Apolipoprotein B levels, transaminases and amma-glutamyl transferase). Oral Glucose Tolerance Test (OGTT) will be performed. The insulin sensitivity and insulin resistance was assessed by calculating HOMA index (Homeostasis Model Assessment) and QUICKI (Quantitative Insulin-Sensitivity Check Index), using the following formulas:

HOMA: fasting plasma insulin in mU/l x FPG in mmol/l/22.5 QUICKI: 1/(log10 fasting plasma insulin in mU/l + log10 glucose in mg/dl)

Inflammatory index (VES, high-sensitive CRP, including fecal calprotectin)

Liver ultrasonography for detection of fatty liver disease

ELIGIBILITY:
Inclusion Criteria:

* 6 <Age <14 years
* Severe obesity (>3 DS) according to WHO classification.
* Gestational age: 37-42 weeks.
* Birth-weight: > 2500 g e < 4000 g
* Caucasian

Exclusion Criteria:

* secondary obesity
* supplementation with pre/probiotics (in the previous 3 months);
* antibiotic treatment (in the previous 3 months);
* chronic or acute intestinal diseases (in the previous 3 months).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota composition. | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on gut microbiota composition and metabolite production. Differences in gut microbiota composition and function will be evaluated in obese children's stools before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months). Study of the microbiota biodiversity will be performed by high-throughput sequencing techniques (16S rRNA gene sequencing) in order to establish whether postbiotics could modulate the microbial composition in obese children
Changes in short-chain fatty acid production by gut microbiota | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on gut microbiota composition and metabolite production. Differences in gut microbiota composition and function will be evaluated in obese children's stools before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months). Analysis of short chain fatty acids concentration by gas-chromatography (GC-FID) will be performed in order to monitor the effect of postbiotics intake modulating microbial metabolite production

SECONDARY OUTCOMES:
Changes in total cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in LDL cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in HDL cholesterol levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in triglycerides levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in fasting glucose levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in fasting insulin levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in HOMA index (Homeostasis Model Assessment) | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in QUICKI (Quantitative Insulin-Sensitivity Check Index) | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in alanine aminotransferase (ALT) levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in aspartate aminotransferase (ALT) levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in gamma glutamyl transferase (GGT) levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in body mass index | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in waist circumference | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in triceps skinfold | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in systemic arterial blood pressure | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Complete cell blood count | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in C-reactive protein (CRP) levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in erythrocyte sedimentation rate (ESR) | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in fecal calprotectin levels | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months).
Changes in body mass composition | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months). body mass composition will be assessed using an air displacement plethysmography system (BOD POD COSMED-USA)
Oral glucose tolerance test (OGTT) result | t0
  Fasting glucose and glucose levels after 2 hours from ingestion of a glucose-containing solution.
Degree of fatty liver disease evaluated by echosonography of the liver | t0: 0 t1: +4 months t2: +8 months
  Interventions aimed at improving diet and lifestyle, on anthropometrics data and glucose and lipid profile before starting the DHA supplementation (t0) and dietary-lifestyle intervention, at the end of DHA supplementation (t1: +4 months) and after 4 months of dietary dietary-lifestyle intervention without DHA supplementation (t2: +8 months). body mass composition will be assessed using an air displacement plethysmography system (BOD POD COSMED-USA)

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Verduci, Study Chair — Hospital San Paolo
Locations (1):
- Ospedale San Paolo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No